CLINICAL TRIAL: NCT06313320
Title: Determination of the Association of Intraoperative Nociception Electroencephalographic Biomarkers and Postoperative Pain
Brief Title: Intraoperative Electroencephalographic Biomarkers of Postoperative Pain
Status: Recruiting | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: OAIC1344-23
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-12

CONDITIONS: Pain Postoperative; Nociceptive Pain
Keywords: Pain; Nociception; Electroencephalogram
MeSH Terms: conditions — Pain, Postoperative; Nociceptive Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — The investigators will collect plasma at 3 timepoints during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to explore whether specific intraoperative EEG signals (brain waves or neuronal electrical activity) are associated with the severity of acute postoperative pain.

DETAILED DESCRIPTION:
This is a prospective minimal-risk observational study to collect and analyze EEG data during intraepidermal electrical stimulation in patients receiving general anesthesia (GA) for abdominal surgery. To collect nociception-related EEG signal during GA the investigators designed a standardized Intraepidermal Electrical Stimulation (IES) Protocol. The intensity of the electrical stimulus will be calibrated to each participant perception pre-surgery, with 3 different intensities: sensitivity threshold, mild-pain threshold, and moderate-pain threshold. The IES will be administered several times throughout the surgical procedure: a) At baseline, prior to induction of GA, b) Three minutes after loss of consciousness, c) Five minutes after fentanyl administration and orotracheal intubation, d) Five minutes after first incision and every 20 minutes until the end of the surgery, and f) After surgery ends and before extubation. To standardize the anesthesia management as much as possible, all patients will be attended by a reduced number of anesthesiologists. The hypnosis will be achieved with propofol, while analgesia will be mainly achieved with either fentanyl or remifentanil. EEG will be recorded with a 32-channel high standard equipment. Once the patient arrives to the Post-Anesthesia Care Unit (PACU), the investigators will record the pain reported by the patient using the Numeric Pain Rating Scale every 15 minutes during the first hour, and every 30 minutes until patient is discharged from the PACU. Also, the investigators will both, record opioid administration through the surgery and estimate their effect-site concentration with pharmacokinetic/pharmacodynamic models. Besides, the investigators will measure opioid plasmatic concentrations.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist Performance Status I or II
* Scheduled for elective laparoscopic abdominal surgery under General Anesthesia

Exclusion Criteria:

* Body Mass Index > 35 kg/m2
* Past history or suspected difficult airway
* Craniofacial malformations
* Use of regional anesthesia technique during or after the surgery
* Severe arrhythmia or use of a pacemaker device
* Severe neuropsychiatric illness (Mayor depression, bipolar disorder, schizophrenia)
* Regular use of psychoactive drugs
* Any injury in the right hand
* Past history of peripheral neuropathy
* Diabetes Mellitus
* Known lesion in the spinothalamic tract.
* Analgesics used in the past 72 hours
* Known allergy to propofol
* Previous diagnosis of a condition associated with chronic pain (such as fibromyalgia, rheumatoid arthritis, osteoarthritis, migraine)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients schedule for elective abdominal surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Pain in PACU | From PACU Admission to PACU Discharged, an average of 2 hours
  Pain is evaluated several times during PACU stay using the Numeric Rating Scale (from 0 to 10). Discrete Numerical Variable

SECONDARY OUTCOMES:
Opioid Consumption in PACU | From PACU Admission to PACU Discharged, an average of 72 hours
  Total opioid administered during PACU stay in Morphine Milligram Equivalent (MME). Continuous Numerical Variable.
Maximum Pain at 24h | From PACU discharged to 24 hours after PACU discharged
  Pain is evaluated several times during hospital stay using the Numeric Rating Scale (from 0 to 10). This outcome corresponds to the maximum pain reported by the patient during the time frame. Discrete Numerical Variable.
Presence of surgical related pain at day 7 | 7 days after the surgery (+- 1 day)
  Pain of any intensity (Numeric Rating Scale >1) reported by the patient 7 days after the surgery
Presence of surgical related pain at day 30 | 30 days after surgery (+- 3 day)
  Pain of any intensity (Numeric Rating Scale >1) reported by the patient 30 days after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Gutierrez, MD, PhD, Principal Investigator — University of Chile
Locations (2):
- Chile (2):
  - Hospital Clinico de la Universidad de Chile, Santiago, RM
  - Centro de Investigacion Clinica Avanzada, Santiago

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Background] Garcia PS, Kreuzer M, Hight D, Sleigh JW. Effects of noxious stimulation on the electroencephalogram during general anaesthesia: a narrative review and approach to analgesic titration. Br J Anaesth. 2021 Feb;126(2):445-457. doi: 10.1016/j.bja.2020.10.036. PMID 33461725
- [Background] Baharloo R, Principe JC, Fillingim RB, Wallace MR, Zou B, Crispen PL, Parvataneni HK, Prieto HA, Machuca TN, Mi X, Hughes SJ, Murad GJA, Rashidi P, Tighe PJ. Slow Dynamics of Acute Postoperative Pain Intensity Time Series Determined via Wavelet Analysis Are Associated With the Risk of Severe Postoperative Day 30 Pain. Anesth Analg. 2021 May 1;132(5):1465-1474. doi: 10.1213/ANE.0000000000005385. PMID 33591118